CLINICAL TRIAL: NCT06136650
Title: MK-5684-004: A Phase 3, Randomized, Open-label Study of Opevesostat Versus Alternative Abiraterone Acetate or Enzalutamide in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) That Progressed On or After Prior Treatment With One Next-generation Hormonal Agent (NHA) (OMAHA-004)
Brief Title: A Study of Opevesostat (MK-5684) Versus Alternative Next-generation Hormonal Agent (NHA) in Metastatic Castration-resistant Prostate Cancer (mCRPC) Post One NHA (MK-5684-004)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5684-004; MK-5684-004 (Other: MSD); jRCT2031240030 (Registry Identifier: Japan Registry of Clinical Trial (jRCT)); 2023-504957-11-00 (Registry Identifier: EU CT); U1111-1288-5002 (Registry Identifier: UTN)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC); Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; fludrocortisone acetate; Hydrocortisone; Abiraterone Acetate; Prednisone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hormone Replacement Therapy (HRT) + Opevesostat (Experimental): Participants receive opevesostat 5 mg by oral tablets twice daily (BID) plus dexamethasone 1.5 mg by oral tablets and fludrocortisone acetate 0.1 mg oral tablet once daily (QD) continuously until disease progression. Hydrocortisone 100 mg (oral or intramuscular [IM]) will also be provided to participants for use as rescue medication.
  Interventions: Drug: Opevesostat; Drug: Dexamethasone; Drug: Fludrocortisone acetate; Drug: Hydrocortisone
- Alternative Next-Generation Hormonal Agent (NHA) (Active Comparator): Participants receive abiraterone 1000mg QD by oral tablets plus prednisone 5 mg BID by oral tablets or enzalutamide 160 mg QD by oral tablets until disease progression.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone acetate; Drug: Enzalutamide

INTERVENTIONS:
Drug: Opevesostat — Administered orally
  Other Names: MK-5684
  Arms: Hormone Replacement Therapy (HRT) + Opevesostat
Drug: Dexamethasone — Administered orally
  Arms: Hormone Replacement Therapy (HRT) + Opevesostat
Drug: Fludrocortisone acetate — Administered orally
  Arms: Hormone Replacement Therapy (HRT) + Opevesostat
Drug: Hydrocortisone — Administered orally or IM as a rescue drug
  Arms: Hormone Replacement Therapy (HRT) + Opevesostat
Drug: Abiraterone acetate — Administered orally
  Other Names: Zytiga; Yonsa
  Arms: Alternative Next-Generation Hormonal Agent (NHA)
Drug: Prednisone acetate — Administered orally
  Arms: Alternative Next-Generation Hormonal Agent (NHA)
Drug: Enzalutamide — Administered orally
  Other Names: Xtandi
  Arms: Alternative Next-Generation Hormonal Agent (NHA)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of opevesostat plus hormone replacement therapy (HRT) compared to alternative abiraterone acetate or enzalutamide in participants with Metastatic Castration-resistant Prostate Cancer (mCRPC) previously treated with one next-generation hormonal agent (NHA). The primary study hypothesis is that opevesostat is superior to alternative abiraterone acetate or enzalutamide with respect to radiographic progression free survival (rPFS) per Prostate Cancer Working Group (PCWG) Modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1), as assessed by Blinded Independent Central Review (BICR), in androgen receptor ligand binding domain (AR LBD) mutation positive and negative participants.

DETAILED DESCRIPTION:
Per Protocol Amendment 08, overall survival (OS) was moved to be a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Have histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while receiving androgen deprivation therapy (ADT) (or post bilateral orchiectomy) within 6 months before screening
* Has current evidence of distant metastatic disease (M1 disease) documented by either bone lesions on bone scan and/or soft tissue disease shown by computed tomography (CT)/magnetic resonance imaging (MRI)
* Has disease that progressed during or after treatment with one next-generation hormonal agent (NHA) for hormone sensitive prostate cancer (HSPC) (metastatic hormone-sensitive prostate cancer [mHSPC] or non-metastatic hormone-sensitive prostate cancer [nmHSPC]), or castration-resistant prostate cancer (CRPC) (metastatic castration-resistant prostate cancer [mCRPC] or non-metastatic castration-resistant prostate cancer [nmCRPC]), for at least 8 weeks of NHA treatment (at least 14 weeks of NHA treatment for participants with bone progression). Note: Participants may have received abiraterone acetate and docetaxel or darolutamide and docetaxel for HSPC. However, participants must have received no more than 6 cycles of docetaxel and had no radiographic disease progression while receiving docetaxel
* Has had prior treatment with poly (ADP-ribose) polymerase inhibitor (PARPi) or were deemed ineligible to receive treatment by the investigator or have refused PARPi treatment
* Has ongoing androgen deprivation therapy (ADT) with serum testosterone <50 ng/dL (<1.7 nM)
* Has an eastern clinical oncology group (ECOG) performance status of 0 or 1 assessed within 10 days before randomization
* Has adequate organ function
* Has provided tumor tissue from a fresh core or excisional biopsy from soft tissue not previously irradiated. Samples from tumors progressing at a prior site of radiation are allowed
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Participants who have adverse event (AEs) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement therapy (HRT) or participants who have ≤Grade 2 neuropathy or ≤Grade 2 osteopenia/osteoporosis are eligible
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has presence of gastrointestinal condition
* Is unable to swallow capsules/tablets
* Has history of pituitary dysfunction
* Has poorly controlled diabetes mellitus
* Has clinically significant abnormal serum potassium or sodium level
* Has any of the following at screening visit: Hypotension: systolic blood pressure (BP) <110 mmHg, or uncontrolled hypertension: systolic BP ≥160mmHg or diastolic blood BP ≥90 mmHg, in 2 out of the 3 recordings with optimized antihypertensive therapy
* Has a history of active or unstable cardio/cerebrovascular disease, including thromboembolic events
* History or family history of long QTc syndrome
* Has a history of seizure(s) within 6 months before providing documented informed consent (IC) or has any condition that may predispose to seizure within 12 months prior to the date of enrollment
* Has a history of clinically significant ventricular arrhythmias or Mobitz II second degree or third-degree heart block without a permanent pacemaker in place
* Has received a taxane-based chemotherapy for metastatic castration-resistant prostate cancer (mCRPC)
* Has not adequately recovered from major surgery or have ongoing surgical complications
* Is currently being treated with Cytochrome P450 (CYP450)-inducing antiepileptic drugs for seizures
* Participants on an unstable dose of thyroid hormone therapy, as judged by the investigator, within 6 months before the start of the study intervention
* Receives prior radiotherapy within 2 weeks before the first dose of study intervention, or radiation-related toxicities, requiring corticosteroids
* Receives prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Has systemic use of strong Cytochrome P450 3A4 (CYP3A4) inducers and P-glycoprotein (P-gp) inhibitors within 2 weeks before the first dose of study intervention
* Has received prior targeted small molecule therapy or NHA treatment within 4 weeks before the first dose of study intervention
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has known hypersensitivity to the components or excipients in abiraterone acetate, prednisone or prednisolone, enzalutamide, fludrocortisone, dexamethasone, or opevesostat
* Has a "superscan" bone scan defined as an intense symmetric activity in the bones and diminished renal parenchymal activity on baseline bone scan such that the presence of additional metastases in the future could not be evaluated
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, (ie, without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during study screening, are clinically stable and have not required steroid treatment for at least 14 days prior to the first dose of study intervention
* Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is allowed
* Active infection requiring systemic therapy
* Has concurrent active Hepatitis B virus and Hepatitis C virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-05-10 (Estimated); Study Completion 2030-12-02 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) | Up to approximately 52 months
  rPFS is defined as the time from randomization to the first documented disease progression per PCWG-modified RECIST 1.1 by BICR or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 82 months
  OS is defined as the time from randomization to death due to any cause.
Time to Initiation of the First Subsequent Anticancer Therapy (TFST) | Up to approximately 82 months
  TFST is defined as the time from randomization to initiation of the first subsequent anti-cancer therapy or death, whichever occurred first.
Objective Response Rate (ORR) | Up to approximately 82 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per PCWG-modified RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Duration of Response (DOR) | Up to approximately 82 months
  For participants who demonstrate confirmed CR or PR, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression per PCWG-modified RECIST 1.1 as assessed by BICR or death from any cause, whichever occurs first.
Time to Pain Progression (TTPP) | Up to approximately 82 months
  TTPP is defined as the time from randomization to pain progression. TTTP is assessed by Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("Worst Pain in 24 Hours") and opiate analgesic use (Analgesic Quantification Algorithm [AQA] Score).
Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G) Total Score | Baseline and up to approximately 82 months
  The FACT-G is a health-related quality of life (HRQoL) 27-item questionnaire in participants being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 (not at all) to 4 (very much). The total score can range from 0 to 108. Higher scores indicate higher HRQoL. The change from baseline in FACT-G total score will be reported.
Time to Deterioration (TTD) in FACT-G Total Score | Up to approximately 82 months
  The FACT-G is a HRQoL 27-item questionnaire in participants being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 (not at all) to 4 (very much). The total score can range from 0 to 108. Higher scores indicate higher HRQoL. TTD in FACT-G total score will be reported.
Overall Improvement in FACT-G Total Score | Up to approximately 82 months
  The FACT-G is a HRQoL 27-item questionnaire in participants being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 (not at all) to 4 (very much). The total score can range from 0 to 108. Higher scores indicate higher HRQoL. The overall improvement in FACT-G total score will be reported.
Time to Prostate-specific Antigen (PSA) Progression | Up to approximately 82 months
  The time to PSA progression is the time from randomization to PSA progression. The PSA progression date is defined as the date of: 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there was PSA decline from baseline; OR 2) ≥25% increase and ≥2 ng/mL increase from baseline.
PSA Response Rate | Up to approximately 82 months
  The PSA response rate is the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by ≥50%. The reduction in PSA level was confirmed by an additional PSA evaluation performed ≥3 weeks from the original response.
Time to First Symptomatic Skeletal-Related Event (TSSRE) | Up to approximately 82 months
  TSSRE is the time from randomization to the first symptomatic skeletal-related event defined as: 1. use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms 2. occurrence of new symptomatic pathologic bone fracture (vertebral or non-vertebral) 3. occurrence of spinal cord compression 4. tumor-related orthopedic surgical intervention, whichever occurs first.
Number of Participants Who Experience an AE | Up to approximately 82 months
  An AE is defined as any unfavorable and unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience one or more AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 82 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (320):
- United States (59):
  - The University of Arizona Cancer Center - North Campus ( Site 0073), Tucson, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 0044), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 0040), Orange, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center (0120), Orange, California
  - Stanford Cancer Center ( Site 0036), Palo Alto, California
  - Emad Ibrahim,MD,INC. ( Site 0012), Redlands, California
  - Kaiser Permanente Riverside Medical Center ( Site 0099), Riverside, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center ( Site 0114), Sacramento, California
  - San Francisco VA Health Care System ( Site 0093), San Francisco, California
  - Kaiser Permanente-Kaiser Permanente, Vallejo Medical Center, Adult Oncology ( Site 0101), Vallejo, California
  - University of Colorado Anschutz Medical Campus ( Site 0046), Aurora, Colorado
  - UCHealth Highlands Ranch Hospital ( Site 0111), Highlands Ranch, Colorado
  - Colorado Clinical Research ( Site 0067), Lakewood, Colorado
  - University of Colorado Health - Lone Tree Medical Center ( Site 0112), Lone Tree, Colorado
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0064), New Haven, Connecticut
  - MedStar Washington Hospital Center ( Site 0103), Washington D.C., District of Columbia
  - Florida Cancer Specialists - South ( Site 7003), Fort Myers, Florida
  - Mount Sinai Cancer Center ( Site 0107), Miami Beach, Florida
  - Memorial Hospital West-Memorial Cancer Institute ( Site 0109), Pembroke Pines, Florida
  - Northside Hospital-Northside Hospital Oncology Network ( Site 0100), Atlanta, Georgia
  - Edward-Elmhurst Healthcare, Elmhurst Hospital-Nancy W. Knowles Cancer Center ( Site 0074), Elmhurst, Illinois
  - Edward-Elmhurst Healthcare, Edward Hospital-Edward Cancer Center ( Site 0075), Naperville, Illinois
  - Illinois Cancer Care ( Site 0104), Peoria, Illinois
  - Urology of Indiana - Carmel ( Site 0055), Carmel, Indiana
  - University of Kentucky Chandler Medical Center ( Site 0048), Lexington, Kentucky
  - Baltimore Veterans Affairs Medical Center ( Site 0069), Baltimore, Maryland
  - Greenebaum Comprehensive Cancer Center ( Site 0049), Baltimore, Maryland
  - Chesapeake Urology ( Site 0009), Towson, Maryland
  - Henry Ford Hospital ( Site 0015), Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 0005), Grand Rapids, Michigan
  - HealthPartners Cancer Research Center-HealthPartners Frauenshuh Cancer Center ( Site 0072), Saint Louis Park, Minnesota
  - HealthPartners Cancer Research Center-HealthPartners Cancer Center at Regions Hospital ( Site 0092), Saint Paul, Minnesota
  - St. Vincent Frontier Cancer Center-Research ( Site 0037), Billings, Montana
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists ( Site 0026), Omaha, Nebraska
  - OptumCare Cancer Care-Research Department ( Site 0078), Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada ( Site 0010), Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey ( Site 0033), New Brunswick, New Jersey
  - Associated Medical Professionals - Urology ( Site 0081), Syracuse, New York
  - University Hospitals Cleveland Medical Center ( Site 0043), Cleveland, Ohio
  - Central Ohio Urology Group - Gahanna ( Site 0098), Gahanna, Ohio
  - Genesis Healthcare System ( Site 0102), Zanesville, Ohio
  - MidLantic urology ( Site 0022), Bala-Cynwyd, Pennsylvania
  - Fox Chase Cancer Center ( Site 0076), Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Health Care System (RHJVAHCS)-Urology ( Site 0083), Charleston, South Carolina
  - Avera Cancer Institute - Pierre ( Site 0118), Pierre, South Dakota
  - Avera Cancer Institute- Research ( Site 0094), Sioux Falls, South Dakota
  - Avera Cancer Institute - Yankton ( Site 0117), Yankton, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 0063), Germantown, Tennessee
  - Texas Oncology - Central/South Texas ( Site 8003), Austin, Texas
  - Texas Oncology - DFW ( Site 8001), Dallas, Texas
  - Texas Oncology - Gulf Coast ( Site 8002), Houston, Texas
  - University of Virginia Health System ( Site 0054), Charlottesville, Virginia
  - Inova Schar Cancer Institute ( Site 0017), Fairfax, Virginia
  - Virginia Cancer Specialists (VCS) ( Site 8004), Fairfax, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0061), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0004), Roanoke, Virginia
  - Spokane Urology ( Site 0035), Spokane, Washington
  - Northwest Cancer Specialists (Compass Oncology) ( Site 8008), Vancouver, Washington
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0020), Milwaukee, Wisconsin
- Australia (5):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0214), Macquarie University, New South Wales
  - Westmead Hospital ( Site 0212), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 0211), Brisbane, Queensland
  - Monash Health ( Site 0219), Clayton, Victoria
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0210), Melbourne, Victoria
- Brazil (14):
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA ( Site 0256), Fortaleza, Ceará
  - Hospital Santa Rita de Cassia ( Site 0271), Vitória, Espírito Santo
  - Obras Sociais Irma Dulce ( Site 0255), Salvador, Estado de Bahia
  - Hospital São Domingos ( Site 0258), São Luís, Maranhão
  - Hospital Mario Penna ( Site 0264), Belo Horizonte, Minas Gerais
  - Universidade Federal do Triangulo Mineiro - Hospital de Clinicas ( Site 0262), Uberaba, Minas Gerais
  - ICTRIALS Pesquisa e Desenvolvimento ( Site 0274), Curitiba, Paraná
  - Hospital Universitário Evangélico Mackenzie ( Site 0252), Curitiba, Paraná
  - Hospital São Lucas da PUCRS ( Site 0270), Porto Alegre, Rio Grande do Sul
  - Clínica de Neoplasias Litoral ( Site 0269), Itajaí, Santa Catarina
  - Hospital Universitário São Francisco de Assis - Bragança Paulista ( Site 0251), Bragança Paulista, São Paulo
  - Hospital de Base de São José do Rio Preto ( Site 0275), São José do Rio Preto, São Paulo
  - Instituto do Câncer Brasil - Unidade Taubaté ( Site 0263), Taubaté, São Paulo
  - Hospital Paulistano ( Site 0259), São Paulo
- Canada (5):
  - Trillium Health Partners - Credit Valley Hospital ( Site 0289), Mississauga, Ontario
  - The Ottawa Hospital - General Campus ( Site 0286), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0285), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0276), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0277), Québec, Quebec
- Chile (6):
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0306), Talca, Maule Region
  - FALP ( Site 0303), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 0304), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0301), Santiago, Region M. de Santiago
  - CIDO SpA-Oncology ( Site 0302), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0305), Viña del Mar, Región de Valparaíso
- China (31):
  - The Second Hospital Of Anhui Medical University ( Site 1633), Hefei, Anhui
  - Peking University First Hospital-Urology ( Site 1602), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Urinary Surgery ( Site 1620), Beijing, Beijing Municipality
  - First Medical Center of Chinese PLA General Hospital ( Site 1601), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 1623), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 1603), Chongqing, Chongqing Municipality
  - Southwest Hospital of Third Military Medical University ( Site 1645), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University-Urology ( Site 1639), Fuzhou, Fujian
  - The first affiliated hospital of Guangzhou medical university ( Site 1637), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center-Urology Surgery ( Site 1638), Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 1632), Wuhan, Hubei
  - The Central Hospital of Wuhan ( Site 1635), Wuhan, Hubei
  - Hubei Cancer Hospital-Urinary surgery ( Site 1631), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 1630), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( Site 1615), Nanjing, Jiangsu
  - Nantong Tumor Hospital-Urology ( Site 1609), Nantong, Jiangsu
  - Wuxi People's Hospital ( Site 1612), Wuxi, Jiangsu
  - The Second Affiliated Hospital of Xi'an Jiaotong University-Oncology Department ( Site 1619), Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology department ( Site 1618), Xi'an, Shaanxi
  - Yantai Yuhuangding Hospital ( Site 1622), Yantai, Shandong
  - Renji Hosp Shanghai Jiaotong U School of Med ( Site 1624), Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University-Urology ( Site 1613), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University-Urology Surgery ( Site 1642), Chengdu, Sichuan
  - Nanchong Central Hospital-urology ( Site 1647), Nanchong, Sichuan
  - The Second Hospital of Tianjin Medical University ( Site 1616), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi-Urology ( Site 1644), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital ( Site 1643), Kunming, Yunnan
  - Zhejiang Provincial People's Hospital-Urology ( Site 1641), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing-urology ( Site 1605), Jiaxing, Zhejiang
  - Ningbo First Hospital-Urology ( Site 1608), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 1604), Wenzhou, Zhejiang
- Colombia (7):
  - Los Cobos Medical Center ( Site 0336), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0326), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0327), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0329), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia ( Site 0328), Piedecuesta, Santander Department
  - Fundación Valle del Lili ( Site 0330), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0334), Cali, Valle del Cauca Department
- Costa Rica (3):
  - CIMCA-Hemato-Oncology ( Site 0380), San José, Provincia de San José
  - Hospital Metropolitano - Sede Lindora-Metropolitano Research Institute Sede Lindora ( Site 0379), Santa Ana, Provincia de San José
  - Onco Tech, S.A. ( Site 0376), San José
- Czechia (6):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0403), Brno, Brno-mesto
  - Krajská nemocnice Liberec-Department of Urology ( Site 0407), Liberec, Liberecký kraj
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 0401), Prague, Praha 5
  - Fakultni Nemocnice u sv. Anny v Brne-Onkologicko-chirurgicke oddeleni ( Site 0404), Brno, South Moravian
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0405), Olomouc
  - Vseobecna fakultni nemocnice v Praze ( Site 0406), Prague
- Estonia (3):
  - East-Tallinn Central Hospital ( Site 1528), Tallinn, Harju
  - North Estonia Medical Centre Foundation ( Site 1526), Tallinn, Harju
  - Tartu University Hospital-Radiotherapy and oncology ( Site 1527), Tartu, Tartu
- France (11):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0451), Strasbourg, Alsace
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 0461), Bordeaux, Aquitaine
  - CENTRE LEON BERARD ( Site 0459), Lyon Cedex08, Auvergne-Rhône-Alpes
  - CHU-BREST Cavale Blanche ( Site 0456), Brest, Finistere
  - Ramsay Santé - Clinical La Croix Du Sud ( Site 0460), Quint-Fonsegrives, Haute-Garonne
  - Centre Bourgogne ( Site 0464), Lille, Hauts-de-France
  - Hôpital Foch ( Site 0455), Suresnes, Hauts-de-Seine
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne ( Site 0454), Clermont-Ferrand, Puy-de-Dome
  - Gustave Roussy ( Site 0452), Villejuif, Val-de-Marne
  - Sainte Catherine Institut du Cancer Avignon Provence ( Site 0458), Avignon, Vaucluse
  - Groupe Hospitalier Paris Saint Joseph ( Site 0465), Paris
- Germany (12):
  - Universitaetsklinikum Freiburg-Klinik für Urologie ( Site 0506), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg ( Site 0531), Heidelberg, Baden-Wurttemberg
  - Studienpraxis Urologie ( Site 0529), Nürtingen, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Site 0521), Munich, Bavaria
  - Caritas-Krankenhaus St. Josef-Klinik fuer Urologie ( Site 0523), Regensburg, Bavaria
  - Universitätsklinikum Marburg-Comprehensive Cancer Center ( Site 0510), Marburg, Hesse
  - Universitätsmedizin Göttingen - Georg-August-Universität-Klinik für Urologie ( Site 0527), Göttingen, Lower Saxony
  - Marien-Krankenhaus ( Site 0515), Bergisch Gladbach, North Rhine-Westphalia
  - Universitaetsklinikum Koeln ( Site 0518), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Urologie ( Site 0528), Dresden, Saxony
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0504), Berlin
  - Vivantes Klinikum Am Urban ( Site 0512), Berlin
- Greece (3):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 0553), Pátrai, Achaia
  - Alexandra General Hospital of Athens-ONCOLOGY DEPT. ( Site 0551), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL-2nd Dep. of Int. Medicine. Research Unit & Diabetes Center ( Site 0552), Chaïdári, Attica
- Guatemala (5):
  - MEDI-K ( Site 0576), Guatemala City
  - CELAN,S.A ( Site 0579), Guatemala City
  - INTEGRA Cancer Institute-Oncology ( Site 0578), Guatemala City
  - Private Practice- Dr. Rixci Augusto Lenin Ramírez ( Site 0577), Guatemala City
  - Sanatorio Nuestra Senora del Pilar ( Site 0580), Guatemala City
- Hong Kong (2):
  - Hong Kong Integrated Oncology Centre ( Site 0603), Central
  - Queen Mary Hospital ( Site 0602), Hong Kong
- Hungary (4):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás C ( Site 0630), Miskolc, Borsod-Abauj Zemplen county
  - Nograd Varmegyei Szent Lazar Korhaz-Onkologia es Sugarterapias Osztaly ( Site 0636), Salgótarján, Nógrád megye
  - Országos Onkológiai Intézet-Urogenitális Tumorok és Klinikai Farmakológiai Osztály ( Site 0631), Budapest, Pest County
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 0632), Debrecen
- Ireland (2):
  - St. Vincent's University Hospital ( Site 0652), Dublin, Dublin
  - Tallaght University Hospital ( Site 0651), Dublin
- Israel (8):
  - Emek Medical Center ( Site 0680), Afula
  - Rambam Health Care Campus-Oncology Division ( Site 0676), Haifa
  - Shaare Zedek Medical Center ( Site 0679), Jerusalem
  - Hadassah Medical Center ( Site 0683), Jerusalem
  - Meir Medical Center. ( Site 0682), Kfar Saba
  - Rabin Medical Center ( Site 0678), Petah Tikva
  - Sheba Medical Center ( Site 0677), Ramat Gan
  - Sourasky Medical Center ( Site 0681), Tel Aviv
- Italy (6):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 1454), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1452), Milan, Lombardy
  - Ospedale Cannizzaro ( Site 1455), Catania
  - Azienda Ospedaliero Universitaria Policlinico Riuniti di Foggia ( Site 1456), Foggia
  - Ospedale San Raffaele-Oncologia Medica ( Site 1451), Milan
  - Azienda Ospedaliera Santa Maria Terni ( Site 1458), Terni
- Japan (30):
  - Toho University Sakura Medical Center ( Site 0730), Sakura, Chiba
  - University of Fukui Hospital ( Site 0735), Eiheiji-cho,Yoshida-gun, Fukui
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 0746), Kitakyushu, Fukuoka
  - Sapporo Medical University Hospital ( Site 0726), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 0756), Sapporo, Hokkaido
  - Kobe University Hospital ( Site 0741), Kobe, Hyōgo
  - Kanazawa Medical University Hospital ( Site 0734), Mukai-awagasaki, Ishikawa-ken
  - Kagawa University Hospital ( Site 0744), Kita, Kagawa-ken
  - Yokohama City University Medical Center ( Site 0733), Yokohama, Kanagawa
  - Mie University Hospital ( Site 0737), Tsu, Mie-ken
  - National Hospital Organization Nagasaki Medical Center ( Site 0748), Ōmura, Nagasaki
  - Nara Medical University Hospital ( Site 0742), Kashihara, Nara
  - Nanbu Tokushukai Hospital ( Site 0755), Shimajiri, Okinawa
  - Kansai Medical University Hospital ( Site 0739), Hirakata, Osaka
  - Bell Land General Hospital ( Site 0740), Sakai, Osaka
  - The University of Osaka Hospital ( Site 0738), Suita, Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 0747), Saga, Saga-ken
  - Nihon University Itabashi Hospital ( Site 0732), Itabashiku, Tokyo
  - The Jikei University Hospital ( Site 0731), Minato, Tokyo
  - Akita University Hospital ( Site 0728), Akita
  - Kyushu University Hospital ( Site 0745), Fukuoka
  - Fukushima Medical University Hospital ( Site 0758), Fukushima
  - Gifu University Hospital ( Site 0736), Gifu
  - Hiroshima University Hospital ( Site 0743), Hiroshima
  - Kagoshima University Hospital ( Site 0754), Kagoshima
  - National Hospital Organization Kumamoto Medical Center ( Site 0749), Kumamoto
  - Miyazaki Prefectural Miyazaki Hospital ( Site 0752), Miyazaki
  - University of Miyazaki Hospital ( Site 0751), Miyazaki
  - Nagano Municipal Hospital ( Site 0757), Nagano
  - National Hospital Organization Oita Medical Center ( Site 0750), Ōita
- Latvia (2):
  - Liepaja Regional Hospital ( Site 1553), Liepāja
  - Pauls Stradins Clinical Univeristy Hospital-Urological department ( Site 1551), Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos ( Site 1576), Kaunas, Kaunas County
  - National Cancer Institute ( Site 1577), Vilnius, Vilniaus Miestas
- Malaysia (5):
  - Hospital Sultan Ismail ( Site 0905), Johor Bahru, Johor
  - University Malaya Medical Centre ( Site 0902), Lembah Pantai, Kuala Lumpur
  - National Cancer Institute ( Site 0904), Putrajaya, Putrajaya
  - Sarawak General Hospital-Radiotherapy Unit ( Site 0901), Kuching, Sarawak
  - Hospital Kuala Lumpur-Radiotherapy and Oncology ( Site 0903), Kuala Lumpur
- Mexico (8):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0928), Guadalajara, Jalisco
  - Health Pharma Professional Research S.A. de C.V: ( Site 0929), Mexico City, Mexico City
  - Higiea Oncologia ( Site 0938), Mexico City, Mexico City
  - Quemex Medical and Research ( Site 0937), Tlalpan, Mexico City
  - Filios Alta Medicina ( Site 0931), Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0932), Monterrey, Nuevo León
  - Eukarya Pharmasite S.C. ( Site 0939), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0934), Oaxaca City, Oaxaca
- New Zealand (2):
  - Dunedin Hospital ( Site 1032), Dunedin, Otago
  - Auckland City Hospital ( Site 1033), Auckland
- Peru (4):
  - Aliada-Oncologìa ( Site 1055), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 1052), Lima
  - Oncosalud-Clinical Research ( Site 1057), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS-Medical Oncology ( Site 1054), Lima
- Portugal (6):
  - Hospital de Cascais Doutor José de Almeida ( Site 1158), Alcabideche, Lisbon District
  - Unidade Local de Saude Gaia/Espinho - Hospital Eduardo Santos Silva ( Site 1156), Vila Nova de Gaia, Porto District
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 1151), Braga
  - Hospital CUF - Tejo ( Site 1157), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 1153), Lisbon
  - Unidade Local de Saude de Santo António - Hospital Santo António ( Site 1152), Porto
- Puerto Rico (3):
  - Advance Urology and Laparoscopic Center ( Site 1178), Ponce
  - Ad-Vance Medical Research-Research ( Site 1177), Ponce
  - Pan American Center for Oncology Trials - Ciudadela ( Site 1176), San Juan
- Romania (4):
  - Spitalul Universitar de Urgență Elias ( Site 1504), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 1503), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 1502), Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie" ( Site 1501), Craiova, Dolj
- Singapore (4):
  - National University Hospital ( Site 1201), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 1202), Singapore, Central Singapore
  - Singapore General Hospital ( Site 1204), Singapore, Central Singapore
  - Tan Tock Seng Hospital-Medical Oncology ( Site 1203), Singapore, Central Singapore
- Slovakia (2):
  - UROEXAM ( Site 1479), Nitra, Nitra Region
  - Privatna Urologicka Ambulancia ( Site 1478), Trenčín, Trenčín Region
- South Africa (6):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE-Clinical Trials Unit ( Site 1230), Port Elizabeth, Eastern Cape
  - Wits Clinical Research ( Site 1234), Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 1232), Pretoria, Gauteng
  - Curo Oncology. ( Site 1237), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 1236), Pretoria, Gauteng
  - Cape Town Oncology Trials ( Site 1233), Cape Town, Western Cape
- South Korea (6):
  - National Cancer Center-Center for Urologic Cancer ( Site 1254), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital-Urology ( Site 1253), Seongnam, Kyonggi-do
  - Kyungpook National University Chilgok Hospital-Urology ( Site 1252), Buk-gu, Kyongsangbuk-do
  - Pusan National University Yangsan Hospital ( Site 1256), Pusan, Kyongsangnam-do
  - Seoul National University Hospital-Urology ( Site 1251), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 1255), Seoul
- Spain (8):
  - Hospital Universitari Parc Tauli-oncologia ( Site 1282), Sabadell, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 1284), Barcelona, Catalonia
  - Institut Català d'Oncologia (ICO) - Girona ( Site 1285), Girona, Gerona
  - Complexo Hospitalario Universitario A Coruna ( Site 1288), A Coruña, La Coruna
  - Hospital Insular de Gran Canaria-Oncology ( Site 1280), Las Palmas de Gran Canaria, Las Palmas
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 1283), Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Burgos-Oncología ( Site 1281), Burgos
  - Hospital Quirón Málaga ( Site 1286), Málaga
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna ( Site 1302), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 1301), Uppsala, Uppsala County
- Taiwan (7):
  - Chi Mei Medical Center ( Site 1336), Tainan, Tainan
  - Kaohsiung Veterans General Hospital ( Site 1337), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 1331), Kaohsiung City
  - China Medical University Hospital-Department of Urology ( Site 1335), Taichung
  - Taichung Veterans General Hospital ( Site 1338), Taichung
  - Taipei Veterans General Hospital ( Site 1332), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Urology ( Site 1334), Taoyuan District
- Thailand (5):
  - Chulalongkorn University ( Site 1355), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1356), Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 1351), Muang, Changwat Khon Kaen
  - Songklanagarind hospital ( Site 1352), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 1353), Muang, Chiang Mai
- Turkey (Türkiye) (9):
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 1379), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1376), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1377), Ankara
  - Koc Universitesi Hastanesi ( Site 1384), Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Baki-Istanbul Bakirkoy Sadi Konuk Training ( Site 1381), Istanbul
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1383), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1378), Istanbul
  - Ege Universitesi Hastanesi-Medical Oncology ( Site 1380), Izmir
  - Samsun Medical Park Hastanesi-medical oncology ( Site 1382), Samsun
- United Kingdom (13):
  - Addenbrooke's Hospital ( Site 1426), Cambridge, Cambridgeshire
  - Royal Derby Hospital ( Site 1431), Derby, Derbyshire
  - Torbay Hospital ( Site 1429), Torquay, Devon
  - Mount Vernon Cancer Centre ( Site 1440), Northwood, England
  - The Royal Cornwall Hospital ( Site 1430), Truro, England
  - The Beatson West of Scotland Cancer Centre ( Site 1428), Glasgow, Glasgow City
  - Charing Cross Hospital-Oncology Research ( Site 1434), London, Hammersmith and Fulham
  - University College London Hospital ( Site 1437), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust-Oncology & Haematology Clinical Trials ( Site 1435), London, London, City of
  - St. George's Hospital-Oncology ( Site 1441), London, London, City of
  - GenesisCare - Oxford ( Site 1442), Oxford, Oxfordshire
  - GenesisCare - Windsor ( Site 1443), Windsor, Windsor And Maidenhead
  - The Christie NHS Foundation Trust ( Site 1436), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26280&tenant=MT_MSD_9011